CLINICAL TRIAL: NCT07309601
Title: Comparison of a Meal Load Between Normal and Functional Variants of the Sucrase-isomaltase (SI) Gene in IBS
Brief Title: Sucrase-Isomaltase (SI) Genes and Meal Load
Acronym: SI IBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Region Skåne FoUU (Unknown)
Responsible Party: Principal Investigator, Bodil Ohlsson, Professor, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-07563-01
Record Dates: First submitted 2025-12-02; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: IBS - Irritable Bowel Syndrome; Sucrase-Isomaltase Deficiency
Keywords: IBS; SI genes; Starch and sucrose; blood glucose levels; bowel symptoms
MeSH Terms: conditions — Irritable Bowel Syndrome; Sucrase-isomaltase deficiency, congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal intake (Experimental)
  Interventions: Dietary Supplement: Meal load

INTERVENTIONS:
Dietary Supplement: Meal load — Meal load during 15 minutes

SUMMARY:
The goal of this interventional study is to examine whether those patients with irritable bowel syndrome (IBS) and a reduced abitility do degrade starch and sugar (lowe levels of enzymes) have lower raise in blood glucose after a meal than those with normal expression of enzymes. We also want to examine whether those IBS patients with reduced enzyme levels have increased bowel symptom in relation to this meal.

The main questions it aims to answer are:

Does reduced ability to degrade starch and sugar due to less enzyme activity lead to lower increase in blood glucose after a meal? Does reduced ability to degrade starch and sugar due to less enzyme activity lead to increased bowel symptoms after a meal?

DETAILED DESCRIPTION:
All IBS patients who have been included in the previous studies (Dnr 2017/171, Dnr 2021-05407-01 and Dnr 2023-01377-01) and have been genetically tested for the sucrase-isomaltse enzyme (SI gene) and other genes encoding enzymes important for carbohydrate absorption will be called and asked if they want to participate in the present study.

The patient receives a basic questionnaire about lifestyle, health and symptoms over the past 2 weeks, including Rome IV questionnaire, irritable bowel syndrome-severity scoring system (IBS-SSS), and visual analog scale for irritable bowel syndrome (VAS-IBS) to be completed at home and brought to the test. The patient comes to the clinic fasting (only allowed to drink water at home in the morning). A plastic tube is placed in the arm, and the patient has to eat a sugar-rich meal during 15 minutes. Blood samples are drawn 10 minutes before start, at the start of the meal, and 10, 20, 30, 45, 60, 90, och 120 minutes aftrewards. Blood samples are analyzed for glucose levels in blood at the Department of Clinical Chemistry, at the hospital. At the same time points as blood sampling, the patient has to complete a questionnaire about bowel symptoms.

Raise in blood glucose and bowel symptoms will be compared between those with reduced enzyme activity and those with normal enzyme activity. The correlation between blood glucose levels and symptoms will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of irritable bowel syndrome (IBS)
* Gene testing has been conducted regarding genes regulating the production of sucrase-isomaltase ensymes in previous dietary interventions using the starch- and sucrose reduced diet (SSRD) or multi-center study.

Exclusion Criteria:

* Diagnosis of inflammatory bowel disease, celiac disease, bile salt malabsorption, gastroenteritis or enteric dysmotility
* Severe food allergy
* Serious heart-, lung-, cardiovascular-, malignant- or mental illness
* Ongoing eating disorder
* Pregnancy
* Recent major gastrointestinal surgery
* Alcohol and/or drug addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes of blood glucose after a meal intake | 2 hours
  We will measure blood glucose levels in plasma through a plastic tube. Two samples will be collected before the meal start. One sample 10 minutes before the meal intake and one immediately prior the meal intake. The meal consists of a sugar-rich breakfast, which must be ingested within 15 minutes. Blood samples will then be collected at 10, 20, 30, 45, 60, 90, and 120 minutes afterwards. Blood glucose will be measured at the Department of Clinical Chemistry at the hospital, according to clinical routines.

SECONDARY OUTCOMES:
Changes of gastrointestinal and extraintestinal symptoms after a meal intake assesssed by self-reported completion on visual analog scales | 2 hours
  The assessment of changes of gastrointestinal and extraintestinal symptoms will be registered during the breakfast meal. The degree of the symptoms abdominal pain; diarrhea; constipation; bloating/flatulence; vomiting/nausea; belching/excess wind; reflux; headache; back pain; muscle/joint pain; and fatigue will be rated by the participants on 100 mm visual analg scales (VAS); one scale for each symptom. 0 mm means no symptoms and 100 means maximal symptoms. The symptoms will be registered at the same tima as the blood samples will be collected. Thus, participants have to register the symptoms 10 minutes before the meal intake, immediately prior the meal intake, and then 10, 20, 30, 45, 60, 90, and 120 minutes afterwards. These VAS scales are extracted from the validated questionnaires the irritable bowel syndrome-severity symptom score (IBS-SSS) and the visual analg scale for irritable bowel syndrome (VAS-IBS).

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Kennbäck, Registered Nurse, Study Chair — Department of Internal Medicine, Skåne University Hospital, 20502 Malmö
Locations (1):
- Skåne University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to ethical rules in Sweden, we can not share individual data. The participants have written an informed concent that data will be presented group wise.